CLINICAL TRIAL: NCT05969600
Title: The Relapses in Childhood Acute Lymphoplastic Leukemia Excluding L3: Experience of Single Institute/ Baghdad
Brief Title: The Relapses in Childhood Acute Lymphoplastic Leukemia Excluding L3
Status: Completed | Type: Observational
Sponsor: Central Teaching Hospital of Peadiatrics, Baghdad (Other)
Responsible Party: Principal Investigator, Maha Kharbat Shadhar Al-Magsoosi, doctor, Central Teaching Hospital of Peadiatrics, Baghdad
Other Study IDs: leukemia
Record Dates: First submitted 2023-06-08; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Leukemia, Acute
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- relapse group
- non-relapse group

SUMMARY:
Background: acute lymphoblastic leukemia is the most common childhood cancer and relapse is the main reason for treatment failure in childhood acute lymphoblastic leukemia.

The aim of this study: is to assess the relapse of childhood acute lymphoblastic leukemia in pediatric patients treated in the Child's Central Teaching Hospital/ Baghdad.

Methods: A retrospective study that reviewed 521 children with newly diagnosed ALL for children below 15 years during the period from 1st of January 2013 to 1st of March 2020 in the hemato-oncology ward in the Child's Central Teaching Hospital in Baghdad, with a total duration of follow-up for two years post last starting treatment (till 1st of March 2022 ).

DETAILED DESCRIPTION:
Six hundred patients diagnosed with acute lymphoblastic leukemia, seventy-nine patients were excluded from study, nine patients died very early before starting induction, seventy patients referred or starting treatment in another centers.

The medical history, laboratory data had been taken for patients including age, gender, residence, date of diagnosis, date of treatment, outcome of induction period and time of relapse, investigations at time of relapse, therapy and relapse outcome were carried out through chart analysis.

The initial diagnosis of ALL was done through bone marrow aspiration morphological classification of blast cells was performed according to the FAB method while immunophenotyping not done for all patients (not available in the period from 2013 to 2016( 227 cases not diagnosed by flowcytometry,294 cases diagnosed by flowcytometry), cytogenetic study not available in our country. The initial diagnostic screen (complete blood count and blood film, renal function test and serum electrolytes and serum uric acid, liver function tests, hepatitis screen, chest x ray, echo-study, computerized tomography and MRI done for indicated cases.

Risk group of patients at time of intial diagnosis divided into standard risk group (age between 1 years and 9.9 years and initial WBC count less than50000) and high risk group (age less than 1 and more than 10 years and WBC count more than 50000 and T cell leukemia) .

Patients regarded and treated as T cell leukemia either by flow cytometry or on clinical bases (mediastinal widening) which associated with(older age,high WBC count, lymphadenopathy, hepatosplenomegaly).

The patients were treated initially with regimens modified from United Kingdom Acute Lymphocytic Leukemia protocols (306 patients were treated by UKALL 2003 for precursor B cell with modification on protocol by increasing the number of intra-thecal dose during period of induction therapy and 22 patients were treated by NHL/BFM 95 protocols for T cell leukemia and used from 1st January 2013 to 1st October 2017, and 193 patients were treated with modified MRC ALL 2011,the modification done by increasing number of intr-thecal dose during the induction period and decreasing high dose of methotrexate from 5 g/m2 to 2g/m2 , from 1st of October to 1st of March 2020) .

The treatment protocols for relapsed cases were modified from MRC-UKALL -R3 protocol , the modification was clofarabin not available and patients were treated by intermediate R3 protocol to adapt local limitation of supportive measures and the shortage of chemotherapeutic agents.

* Infantile leukemia was treated with same protocol and treated as high risk group.
* CNS positive at time of patients presentation treated according to their age and WBCs count .
* Limitation of study : cytogenetic study and MRD are not available in country at time of study .
* B.M.A was done at day eight and day fifteen after started induction and according to the results shifted to another protocol.

Definition of relapse:

An isolated BM relapse was diagnosed with 25% lymphoblast in the BM and without evidence of leukemia at extra medullary sites. Accordingly, isolated extramedullary relapses were those with the clinically-overt extramedullary manifestation of leukemia and less than 5% marrow infiltration. CNS relapse was diagnosed in the case of positive the unequivocal presence of lymphoblasts per microliter CSF or clinical signs of CNS leukemia such as facial nerve palsy, brain/eye involvement .

Testicular relapse was diagnosed by clinical examination and ultrasound, the involvement of any other extramedullary site was confirmed histologically.in this study one case presented with late relapse of cervical lymph node and biopsy done that show T lymphoblastic lymphoma with blast cell less than 1% in B.M. In children with proven leukemia at extramedullary sites, a combined relapse was diagnosed with marrow involvement of lymphoblasts.

Complete remission was defined as the absence of leukemic blasts in peripheral blood and CSF and less than 5% blast on bone marrow aspirate smear, together with hematopoietic regeneration and no evidence of extramedullary (localized) disease.

Induction failure was defined as the failure to achieve remission after 1 month of therapy.

Abandonment of treatment was defined as care termination by the parent/caregiver and/or if more than 4 weeks was exceeded with a no-show/non-attendance for a scheduled treatment by the patient .

Overall survival defined as the time from date of diagnosis and or start treatment to the date of death.

Time of relapse

Based on time factor, relapses were categorized as:

* Very early: within 18 months of diagnosis, while on chemotherapy
* Early: occurred after 18 months of diagnosis and within 6 months of treatment completion
* Late: relapse documented more than 6 months after completion of therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with acute lymphoplastic leukemia

Exclusion Criteria:

* patients died before starting induction chemotherapy.
* patients referred to another oncological center.
* those who starting the treatment in another oncological center

Ages: 2 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A retrospective study that reviewed 521 children with newly diagnosed ALL for children below 15 years during the period from 1st of January 2013 to 1st of March 2020 in the hemato-oncology ward in the Child's Central Teaching Hospital in Baghdad, with a total duration of follow-up for two years post last starting treatment (till 1st of March 2022 ).
Sampling Method: Non-Probability Sample
Enrollment: 521 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
the relapse of childhood acute lymphoblastic leukemia in pediatric patients treated in the Child's Central Teaching Hospital/ Baghdad | the period from 1st of January 2013 to 1st of March 2020
  521 children reviewed with newly diagnosed ALL for children below 15 years

IPD SHARING:
Plan to Share IPD: Undecided